CLINICAL TRIAL: NCT02037750
Title: Foster Teens' Risk During Transition: Preventing Drug Use, HIV, & School Problems
Brief Title: Foster Teens' Risk During Transition
Acronym: LINKS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Social Learning Center (Other)
Collaborators: San Diego State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01DA032634 (NIH)
Record Dates: First submitted 2014-01-13; First posted 2014-01-16 (Estimated); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: School Adjustment; Foster Care Disruptions
Keywords: foster care; school adjustment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LINKS (Experimental): Foster parent and child participate in 16-week intervention
  Interventions: Behavioral: LINKS
- Services as Usual (No Intervention): Foster parent and child receive standard services through child welfare system

INTERVENTIONS:
Behavioral: LINKS — In the LINKS, foster/kin parents will participate in weekly group meetings led by well-trained and supervised paraprofessional facilitators (school behavioral aids and foster parents) where the curriculum is based on parent management training (PMT). In previous studies, attendance at such groups has been high, averaging about 75-80%. Missed sessions will be "made up" with an in-person visit to the foster/kin home during the week of the original session. In addition, youth in the intervention condition will receive individual skill building sessions from a Life Skills Coach to increase their competency at goal setting, refusal skills, and peer relations.
  Arms: LINKS

SUMMARY:
The purpose of this study is to conduct a randomized effectiveness trial to determine whether adding a preventive intervention at the transition from elementary to middle school is effective and cost effective in terms of ameliorating outcomes such as drug and tobacco use, participation in HIV- risking sexual behavior, delinquency, mental health problems, and school failure for young adolescents in foster care. The proposed LINKS intervention marries the goals of child welfare and educational systems. The aims are: a) to determine the effectiveness of the LINKS intervention on key behavioral health and school adjustment outcomes, b) to examine mechanisms of action; specifically the mediating effects of placement failure on outcomes, c) to examine the moderating role of fidelity on outcomes, and d) to examine cost effectiveness and cost avoidance of LINKS.

ELIGIBILITY:
Inclusion Criteria:

* the focal youth will be transitioning into middle school
* the focal youth is in either a foster or kinship care home
* the focal youth has been in the home for a minimum of 30 days (including those who are newly placed in care and those moving from another type of placement).

Exclusion Criteria:

* youth who are are considered medically fragile (i.e., severely physically or mentally handicapped)

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 173 (Actual)
Dates: Start 2012-12; Primary Completion 2018-06 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Number of Placement Failures | between Baseline and 18-Months later

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Chamberlain, Phd, Principal Investigator — Oregon Social Learning Center
Locations (2):
- United States (2):
  - San Diego State University Foundation, San Diego, California
  - Oregon Social Learning Center, Eugene, Oregon